CLINICAL TRIAL: NCT05842044
Title: NSAID Use After Robotic Partial Nephrectomy (No-PAIN): a Randomized, Controlled Trial
Brief Title: NSAID Use After Robotic Partial Nephrectomy
Acronym: No-PAIN
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Mark L. Gonzalgo, MD, PhD, Professor of Clinical, University of Miami
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20220783
Record Dates: First submitted 2023-04-24; First posted 2023-05-03 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-09

CONDITIONS: Kidney Cancer; Renal Cancer; Renal Neoplasm
Keywords: Non-steroidal anti-inflammatory drugs (NSAIDs)
MeSH Terms: conditions — Kidney Neoplasms | interventions — Ketorolac; Ketorolac Tromethamine; Acetaminophen; Oxycodone; Hydromorphone; Ibuprofen

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Masking Description: After study recruitment, the patient will be randomized to the NSAID group (group 1) vs. the no-NSAID group (group 2). Randomization will be masked until after the renorrhaphy is completed and the surgical team will administer versus not administer ketorolac based on group assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1: NSAID (Experimental): Participants in this group will be prescribed NSAIDs instead of the standard of care treatment. Participants will be in this group for approximately 21 days.
  Interventions: Drug: Ketorolac; Drug: Acetaminophen; Drug: Oxycodone; Drug: Hydromorphone; Drug: Ibuprofen
- Group 2: No-NSAID (Active Comparator): Participants in this group will follow standard of care treatment. Participants will be in this group for approximately 21 days.
  Interventions: Drug: Acetaminophen; Drug: Oxycodone; Drug: Hydromorphone

INTERVENTIONS:
Drug: Ketorolac — 15-30mg Ketorolac administered via injection during intraoperative period every six (6) hours during post-surgery (inpatient) period.
  Other Names: Ketorolac tromethamine; Toradol; Biorolac
  Arms: Group 1: NSAID
Drug: Acetaminophen — 1000mg Acetaminophen administered orally during preoperative period. Standardized regimen of Acetaminophen administered during post-surgery (inpatient) period, during postoperative follow-up period.
  Other Names: Tylenol
Drug: Oxycodone — Standardized regimen of Oxycodone administered orally (PO) on demand for moderate pain during post-surgery (inpatient) period.
  At discharge 5mg Oxycodone will be administered to participants on demand if pain score is greater than 7, or if participant required greater than 25mg Oxycodone during the hospitalization.
  Other Names: Oxycontin; Roxicodone
Drug: Hydromorphone — Standardized regimen of Hydromorphone administered intravenously (IV) on demand for severe pain during post-surgery (inpatient) period.
  Other Names: Dihydromorphinone; Dilaudid; Hydromorph Contin; Palladone
Drug: Ibuprofen — 400mg Ibuprofen tablets administered orally (PO) every eight (8) hours for 5 days.
  Other Names: Advil; Motrin
  Arms: Group 1: NSAID

SUMMARY:
The purpose of this study is to see how effective non-steroidal anti-inflammatory drugs (NSAIDs) are at controlling pain without side effects in participants after robotic-assisted partial nephrectomy.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing uncomplicated robotic assisted laparoscopic partial nephrectomy for renal mass at the University of Miami Hospital and Network Sites (Deerfield Beach, Plantation, Lennar (Coral Gables), and Kendal).
* Age 18-99.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Allergy to NSAIDs
* Myocardial infarction or unstable angina within 12 months.
* Any history of coronary artery bypass graft surgery.
* History or active peptic ulcer disease, gastrointestinal (GI) bleeding, GI perforation. History of bleeding disorder. Glomerular filtration rate (GFR) < 60 mL/min/1.73m2 (Modification of Diet in Renal Disease (MDRD) equation).
* Taking any anti-platelet or anti-coagulation medications concurrently (e.g. warfarin, aspirin, clopidogrel, rivaroxaban etc.)
* Chronic opioid use (use within 12 weeks) or history of opioid use disorder.
* Solitary kidney.
* Pregnancy.
* Inability to give informed consent or unable to meet requirement of the study for any reason.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2023-09-15 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Rate of Opioid Use in Postoperative Period | Up to 20 days
  Rate of opioid use is defined as the number of participants who used opioid medications during the post-operative period (defined as end of surgery to post-operative follow up visit) divided by total number of participants in the group at postoperative visit.

SECONDARY OUTCOMES:
Rate of Opioid Medication Use during Hospitalization | Up to 24 hours
  Rate of opioid medication use among study participants during hospitalization, defined as the number of participants who use opioid medication divided by total number of participants in the group during the time between surgery and discharge.
Pain Score Assessed by Standardized Script | Up to 20 days
  At 24 hours post-surgery and during the postoperative follow-up period, pain score will be elicited from study participants using a standardized script, and scored on scale of 0 to 10, with 0 being no pain and 10 being the worst pain.
Pain Score Assessed by International Pain Outcome Questionnaire | Up to 20 days
  Participants will complete the International Pain Outcome questionnaire during the postoperative and follow-up periods. Scores range from 0 to 10, with higher scores indicating more pain.
Number of Treatment-Related Adverse Events | Up to 20 days
  The number of treatment-related of adverse events among study participants will be assessed by treating physician, post-surgery and after discharge during the postoperative period.
Change in Rate of Acute Kidney Injury | Baseline, Up to 20 days
  Rate of acute kidney injury at postoperative follow-up visit. Acute kidney injury is defined as a rise of Creatinine greater than (>) 0.3 from baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Mark L Gonzalgo, MD, PhD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No